CLINICAL TRIAL: NCT04881409
Title: Nasal High-flow Compared to Non-invasive Ventilation in Treatment of Acute Acidotic Hypercapnic Exacerbation of Chronic Obstructive Pulmonary Disease - a Randomized Controlled Noninferiority Trial
Brief Title: Nasal High-flow Compared to Non-invasive Ventilation in Treatment of Acute Acidotic Hypercapnic Exacerbation of Chronic Obstructive Pulmonary Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Hubert Wirtz, Head of Pneumology, University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ELVIS
Record Dates: First submitted 2021-04-28; First posted 2021-05-11 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: COPD Exacerbation Acute
Keywords: nasal high-flow; non-invasive ventilation
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: randomization to NHF or NIV
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nasal high-flow (Experimental): Patient with AECOPD is treated with NHF.
  Interventions: Device: Respiratory support with nasal high-flow (NHF)
- non-invasive ventilation (Active Comparator): Patient with AECOPD is treated with NIV
  Interventions: Device: Respiratory support with non-invasive ventilation (NIV)

INTERVENTIONS:
Device: Respiratory support with nasal high-flow (NHF) — Patient with AECOPD is treated with NHF.
  Arms: nasal high-flow
Device: Respiratory support with non-invasive ventilation (NIV) — Patient with AECOPD is treated with NIV.
  Arms: non-invasive ventilation

SUMMARY:
The ELVIS study compares the nasal high-flow to non-invasive ventilation in treatment of acute acidotic hypercapnic exacerbation of chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
The ELVIS study is a prospective, randomized, multi-centre open label trial following a non-inferiority design to compare the nasal high-flow (NHF) to non-invasive ventilation (NIV) in treatment of acute acidotic hypercapnic exacerbation of chronic obstructive pulmonary disease. Accoring to the randomization the patient is treated with NHF or NIV until discharge. A change of device is possible, if switch criteria are fulfiled OR need for intubation criteria are met before 72h (timepoint for primary endpoint).

ELIGIBILITY:
Inclusion Criteria:

1. acute hypercapnic exacerbation of chronic obstructive pulmonary disease with pH < 7.35
2. pCO2 > 45mmHg
3. age ≥ 18 years
4. written informed consent

Exclusion Criteria:

1. immediate need for intubation (acc. to intubation criteria in this protocol)
2. pH < 7.15
3. BMI ≥ 35 kg/m²
4. established home-NIV or home-CPAP
5. end-stage disease with DNI/DNR order
6. diseases that could influence the primary endpoint: e.g. acute heart infarction, cardiogenic lung edema, acute and massive lung embolism (hypertensive), chronic dialysis with metabolic acidosis, unstable rib fracture influencing ventilation, injury to the face prohibiting use of a face mask
7. acute disease that precludes participation in the trial
8. tracheotomized patients
9. psychological/mental or other inabilities to supply required informed consent
10. participation in other interventional trials
11. suspected lack of compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2021-05-06 (Actual); Primary Completion 2024-02-06 (Estimated); Study Completion 2024-10-06 (Estimated)

PRIMARY OUTCOMES:
Proportion with treatment failure of allocated respiratory support within 72 h after start of respiratory support. | start of treatment until 72 hours
  Treatment failure defined as
  1. intubation or
  2. switch to another method of non-invasive ventilation or
  3. death

SECONDARY OUTCOMES:
intubation within 72 hours (component of primary outcome) | start of treatment until 72 hours
  independent of whether or not responsible primary endpoint
proportion intubated within 7 calendar days after hospitalisation/randomization | start of treatment until 7 calender days after hospitalisation/randomization
Overall survival at day 28 and day 90 | start of treatment until day 90 after start of treatment
(Invasive) ventilator-free days until day 28 | start of treatment until day 28 after start of treatment
(Invasive) ventilator-free hours until the primary endpoint is reached or 72 hours, whichever comes first | start of treatment until maximum 72 hours after start of treatment
Intensive care unit (ICU) and hospital lengths of stay | start of treatment until discharge or day 90 after start of treatment (whichever comes first)
Proportion requiring sedation | start of treatment until discharge or day 90 after start of treatment (whichever comes first)
switch to another method of non-invasive ventilation within 72 hours (component of primary outcome) | start of treatment until 72 hours
  independent of whether or not responsible primary endpoint
death within 72 hours (component of primary outcome) | start of treatment until 72 hours
  independent of whether or not responsible primary endpoint

CONTACTS AND LOCATIONS:
Locations (6):
- Germany (6):
  - München-Klinik Bogenhausen, München, Bavaria
  - Klinikum Emden, Emden, Lower Saxony
  - Lungenklinik Hemer, Hemer, North Rhine-Westphalia
  - University Hospital Leipzig, Leipzig, Saxony
  - Sana Kliniken Ostholstein, Oldenburg in Holstein, Schleswig-Holstein
  - Evangelische Lungenklinik, Berlin

IPD SHARING:
Plan to Share IPD: Yes
According to the recommendations on data sharing by the International Committee of Medical Journal Editors (ICMJE) data resulting from the ELVIS trial will be made available to the scientific community.
Supporting Information: Study Protocol, SAP
Time Frame: After publication of the major results
Access Criteria: After publication of the major results and upon reasonable request from researchers performing an individual patient data meta-analysis, individual patient data that underlie published results will be shared after de-identification. This requires approval by the local ethics committee of the researcher requesting the data along with public registration of the meta-analysis. The coordinating investigator will contact the data protection officer before de-identification to ensure a correct and actual implementation of this process.
  Summary statistics that go beyond the scope of published material will be made available to researchers for meta-analysis upon reasonable request and if the necessary data analysis is not unduly time-consuming. Together with publication of the main results, the trial protocol in full will be made publically available as well as the statistical analysis plan.

REFERENCES:
- [Derived] Braunlich J, Koppe-Bauernfeind N, Petroff D, Franke A, Wirtz H. Nasal high-flow compared to non-invasive ventilation in treatment of acute acidotic hypercapnic exacerbation of chronic obstructive pulmonary disease-protocol for a randomized controlled noninferiority trial (ELVIS). Trials. 2022 Jan 10;23(1):28. doi: 10.1186/s13063-021-05978-z. PMID 35012620

DOCUMENTS (1):
  • Study Protocol (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/09/NCT04881409/Prot_000.pdf